CLINICAL TRIAL: NCT02608307
Title: Adolescent and Young Adult, Parental, and Health Care Provider Decision Making Using Conjoint Analysis
Brief Title: Medical Treatment Decision Making Using Adaptive Conjoint Analysis
Status: Terminated | Type: Observational
Why Stopped: Slow accrual and COVID-19 restrictions
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AYACA
Record Dates: First submitted 2015-11-13; First posted 2015-11-18 (Estimated); Last update posted 2021-12-21 (Actual); Status verified 2021-10

CONDITIONS: Cancer; Brain Tumor; Solid Tumor; Leukemia; Lymphoma
Keywords: Treatment Decision-Making; Adolescents and Young Adult Oncology
MeSH Terms: conditions — Neoplasms; Brain Neoplasms; Leukemia; Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- AYA patients: Adolescence and young adults (AYA) who meet eligibility criteria and consent to participate in the study.
- Parents of AYA patients: Parents of AYA patients who meet eligibility criteria and consent to participate in the study.
- Health Care Providers (HCPs): Health care providers who meet eligibility criteria and consent to participate in the study.

SUMMARY:
In the setting of progressive or recurrent cancer, adolescent and young adult (AYA) patients, parents, and healthcare providers (HCP) are faced with multiple therapeutic options. Each treatment option has a unique risk/benefit ratio, resulting in a need to trade one desirable outcome for another or accept acute toxicities and treatment-related morbidity to increase the chance of survival. Adding to the complexity of this decision, stake holders characterize and value the risk/benefit ratios differently.

This study seeks to learn what things are important to an adolescent or young adult with cancer, parents, and health care providers when making decisions about their treatment choices.

PRIMARY OBJECTIVE: To quantify the relative importance of various factors believed to be important to adolescent and young adult patients with cancer, parents, and health care providers when choosing between treatment options in the hypothetical situation of progressive or refractory disease.

DETAILED DESCRIPTION:
Data for this observational study will be collected first at the time the participants enroll in the study. If the participant agrees to be re-contacted in the event of disease relapse or recurrent cancer, follow-up data will be collected at a second time point up to five years after enrollment. This second follow-up time point is optional.

Participants will complete two short questionnaires and a guided survey on a laptop computer. AYA patients and parents will participate in an interviewer-led interview session. The surveys are the Herth Hope Index (HHI) to assess hope in adults in clinical settings, and the Decision Making Preference Questionnaire (DMPQ) to identify factors that parents believe influence their role in treatment decision making. The guided survey presents a hypothetical situation outlining different treatment options at the time of recurrent or progressive disease. Participants will be asked to answer questions related to type of treatment, location of treatment, hospital of treatment, route of treatment, symptoms or side effects from treatment, quality of life, frequency of clinic visits, chance of being hospitalized, chance of cure, and survival length of time.

Medical data including cancer diagnosis, date of diagnosis, duration of time on treatment, and serious side effects and complications of treatment will be collected on AYA patients.

Data will be analyzed by group: (1) adolescent and young adult patients, (2) parents, or (3) health-care providers.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be English speaking.
* There are three main participant subsets for the first time point of the study:

  * AYA patients (aged 13-30) with an oncological diagnosis who are currently receiving active treatment at St. Jude Children's Research Hospital that includes at least chemotherapy, and have been doing so for at least one month or who completed treatment (that includes at least chemotherapy) less than 1 month prior to enrollment.
  * Parents of a patient (<18) who meets the above criteria. If available, parents of a young adult patient (≥18) who meets the above criteria will be invited to participate.
  * HCPs of patients at St. Jude with at least 1 year of experience taking care of AYA oncology patients. HCPs must have an MD or DO degree and be an attending physician or clinical fellow at St. Jude Children's Research Hospital.
* Patient participants must have an oncological diagnosis that confers less than a 75% overall survival based on consultation with an oncologist.
* Participants who agree to be re-contacted up to five years later, to consider taking part in the T2 time point, must have participated in the T1 time point and the patient participant must have relapsed or recurrent disease at the time of re- contact, as documented in the medical record.

Exclusion Criteria:

* Patients with relapsed or recurrent disease at the time of initial enrollment.
* Patients who only receive local radiation for treatment without adjunctive chemotherapy.
* Patients or parents who are unable to complete the study due to ill health, cognitive compromise, or concern about potential distress based on consultation with a psychosocial provider.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be patients at St. Jude Children's Research Hospital, their parents and health-care providers who consent to enroll in the study. All participants must meet inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2016-02-09 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2019-10-17 (Actual)

PRIMARY OUTCOMES:
Part Worths | Once at participant enrollment
  Conjoint analysis picks a small subset of possible answer combinations and combination sets and asks respondents which option (profile) they prefer in each set. This data is compiled and a hierarchical Bayesian approach, as implanted in Sawtooth Software package, is used to evaluate the relationship between various attributes and the decision choice. The relative importance of various factors on the decision-making process will be evaluated for three groups (patients, parents and HCPs) independently, generating three separate models. At completion of the survey, the part worth for each different treatment attribute (type, location, hospital, route, symptoms or side effects, frequency of clinic visits, chance of hospitalization, quality of life, chance of cure, and survival length of time) is calculated. They are analyzed simultaneously for each participant and only have meaning in relation to one another constituting a single primary outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Blazin, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols